CLINICAL TRIAL: NCT00571753
Title: A Double-blind, Multicentre, Parallel Group, Randomised, Controlled Trial to Evaluate the Possible Benefit of Isoniazid Dose Adjustment According to the Genotype for NAT2 (Arylamine N-acetyltransferase Type 2) in Patients With Pulmonary Tuberculosis
Brief Title: Isoniazid Dose Adjustment According to NAT2 Genotype (IDANAT2)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrolling participants has halted prematurely due to a low recruitment rate.
Sponsor: University of Cologne (Other)
Responsible Party: University of Cologne, Sponsor representative: Prof. Dr. med. Uwe Fuhr, Institute of Pharmacology, University Hospital, University of Cologne, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IDANAT2; EUDRACT Number:2007-000224-41
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-02

CONDITIONS: Pulmonary Tuberculosis
Keywords: pulmonary tuberculosis; NAT2 genotyping; hepatotoxicity of isoniazid
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Isoniazid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test (Experimental): Isoniazid dose adapted according to NAT2 status i.e. appr. 2.5 mg/kg, 5 mg/kg and 7.5 mg/kg for slow, intermediate and rapid acetylators, respectively
  Interventions: Drug: isoniazid
- Control (Active Comparator): Treatment with standard isoniazid dose (appr. 5 mg/kg b.w.)
  Interventions: Drug: isoniazid

INTERVENTIONS:
Drug: isoniazid — modified daily isoniazid dose according to NAT2 genotype (appr. 2.5 mg/kg, 5 mg/kg and 7.5 mg/kg for slow, intermediate and rapid acetylators, respectively).
  Arms: Test
Drug: isoniazid — Treatment with a standard isoniazid dose of isoniazid (appr. 5 mg/kg b.w.)
  Arms: Control

SUMMARY:
The study is conducted to compare safety and efficacy of isoniazid administered as an adjusted dose based on NAT2 (arylamine N-acetyltransferase type 2)genotype and as a standard dose.

The hypothesis is that the genotype-adjusted dose is superior to the standard dose with regard to hepatotoxicity and early treatment failure, respectively, in the group of slow and rapid acetylators of NAT2.

ELIGIBILITY:
Inclusion Criteria:

* Patient is informed and given ample time and opportunity to think about her/his participation and has given her/his written informed consent
* Patient is willing and able to comply with all trial requirements, inclusive genotyping procedure
* Patient is between 18 and 75 years of age (inclusive) during the whole trial, male or female
* Patient has newly diagnosed pulmonary tuberculosis for whom daily antituberculosis therapy is indicated
* Patient has a smear-positive sputum
* Patient has radiological evidence of a pulmonary infiltrate.

Exclusion Criteria:

* Patients with known contraindications for isoniazid: acute hepatitis, macroscopic hematuria, allergy to isoniazid, peripheral neuritis, coagulopathy, severe haemorrhagic diathesis, seizure disorders, psychosis
* Patients with advanced or unstable chronic liver disease which is confirmed on results of biochemical or serological tests by eligibility assessment (relevant abnormalities of the following liver tests: ALT, AST, AP, total and conjugated bilirubin; positive serology for hepatitis), if the assessed risk-benefit ratio for the participation in the study is unfavourable (inclusion upon a decision of clinical investigator)
* Patients with a severe, life-threatening disease with a life expectancy of less than 2 years
* Patients known to have AIDS (CD4+ count <200/ml) or HIV-seropositive patients who are receiving HAART (highly active antiretroviral therapy). Note: HIV-positive patients may be included
* Patients with diabetes mellitus
* Patients with renal insufficiency (creatinine clearance < 30mL / min / 1.73m2) and patients on hemodialysis
* Patients with any other clinical conditions suggesting that he/she should not be included (decision of the clinical investigator)
* Patients with chronic infections requiring concomitant systemic antibacterial agents that are also active against M. tuberculosis (i.e. fluoroquinolones, aminoglycosides, macrolides)
* Patients with intake of systemic antibacterial agents that are also active against M. tuberculosis (i.e. fluoroquinolones, aminoglycosides, macrolides) within 4 weeks prior to antituberculosis treatment
* Patients who have ever received antituberculosis chemotherapy
* Patients who take any hepatotoxic agent on regular basis or have taken it within 3 month before study onset
* Patients with known drug / continuous severe alcohol abuse (drinking more than 60 g alcohol daily)
* Patients who participate in other interventional clinical studies;
* Female patients who are pregnant or lactating;
* Female patients not willing and capable to use two different contraceptive methods throughout the study, e.g. double barrier methods (e.g. diaphragm and condom by the partner, intrauterine devise and condom, sponge and condom, spermicide and condom). Acceptable alternatives of effective contraception are also sexual abstinence or vasectomized partner. In contrast, oral contraceptives are not recommended, since the effectiveness of them may be reduced due to a possible interaction with rifampicin
* Patients who are placed in a closed institution as a result of a court or any other authorities' decision
* Patients who are known or suspected not to comply with the study directives and/or known or suspected not to be reliable or trustworthy
* Patients who are known or suspected not to be capable of understanding and evaluating the information that is given to them as part of the formal information policy (informed consent), in particular regarding the foreseeable risks to which they will be exposed.
* Patients with any of followings will not be included into evaluation for efficacy:

  * Infection with Mycobacterium avium complex
  * Resistance of M. tuberculosis to isoniazid at the first screening test (initial culture).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-12 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of early treatment failure, defined as continuous or recurrently positive sputum cultures | occurring up to week 8 of therapy

SECONDARY OUTCOMES:
Further adverse events of isoniazid | up to week 8 of therapy
Time course of sputum conversion | up to week 8 of therapy
Duration of hospitalization | up to week 8 of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Fätkenheuer, Prof. Dr. med., Principal Investigator — Department I of Internal MedicineUniversity Hospital, University of Cologne
Locations (12):
- Specialized Hospital for Active Treatment of Pulmonary Diseases "Sveta Sofia", Sofia, Bulgaria
- Germany (9):
  - Zentralkrankenhaus Bad Berka GmbH, Bad Berka
  - Karl-Hansen-Klinik, Bad Lippspringe
  - Helios Klinikum Emil von Behring GmbH, Berlin
  - Department I of Internal Medicine, University Hospital, University of Cologne, Cologne
  - Medizinische Klinik I, Abteilung Pneumologie/Allergologie, Universitätsklinikum Frankfurt am Main, Frankfurt am Main
  - Abteilung Innere Medizin/ Pneumologie, Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg
  - Lungenfachklinik Immenhausen, Immenhausen
  - Diakoniekrankenhaus Rotenburg, Rotenburg (Wümme)
  - Division of Infectious Diseases and Clinical Immunology, Department of Internal Medicine, Ulm
- Poland (2):
  - Specialized Hospital of Lung Diseases and Tuberculosis in Wielkopolska in Chodzież, Chodzież
  - Department of Pulmonal Diseases, K. Marcinkowski University of Medical Sciences, Poznan